CLINICAL TRIAL: NCT00665756
Title: Comparison of Efficacy Between Silicone Ahmed Glaucoma Valves and Second Trabeculectomy in Glaucoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Augusto Paranhos Jr, PHD, Federal University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLAU0037
Record Dates: First submitted 2008-04-23; First posted 2008-04-24 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Open Angle Glaucoma
Keywords: Glaucoma; Drainage implant; Ahmed valve; Second trabeculectomy
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma | interventions — Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): second trabeculectomy
  Interventions: Procedure: second Trabeculectomy
- 2 (Active Comparator): Ahmed silicone drainage device implantation
  Interventions: Procedure: Ahmed Implant

INTERVENTIONS:
Procedure: second Trabeculectomy — second trabeculectomy with mitomycin-c
  Other Names: re-Trabeculectomy with mitomycin-C
  Arms: 1
Procedure: Ahmed Implant — Ahmed silicone drainage device
  Other Names: Armed FP-7 adult silicone valve
  Arms: 2

SUMMARY:
In the management of open angle glaucoma, frequently more then one procedure is necessary to control the intra ocular pressure. There is still no consensus whether this second intervention should be a second trabeculectomy or a shunt device. In the present study we compare a second trabeculectomy versus Ahmed silicone shunt device in open angle glaucoma patients with previous trabeculectomy without proper IOP control.

DETAILED DESCRIPTION:
In the management of open angle glaucoma, frequently more then one procedure is necessary to control the intra ocular pressure. There is still no consensus whether this second intervention should be a second trabeculectomy or a shunt device. In the present study we compare a second trabeculectomy versus Ahmed silicone shunt device in open angle glaucoma patients with previous trabeculectomy without proper IOP control.

40 Patients with clinically uncontrolled open angle glaucoma with previous trabeculectomy surgery were selected from the glaucoma sector of Federal university of Sao Paulo. Patients were randomized to one of two groups:

1. Silicone Ahmed Implant
2. Second trabeculectomy

Surgery description:

Ahmed silicone tube implant: A fornix-based conjunctival flap was created between two adjacent recti muscles. Before placement of the tube implant body to the sclera, tube was irrigated with saline solution to open the valve mechanism. The implant's polypropylene body was sutured to sclera with 6.0 silk suture. The tube then trimmed and the anterior chamber was entered from 1mm posterior to corneoscleral limbus with 23-gauge needle. A human donor scleral flap was placed over the tube and sutured to the sclera with 10.0 nylon suture. The conjunctiva was sutured to the limbus.

Second Trabeculectomy: A fornix-based conjunctival flap was created in the opposite superior quadrant of the previous trabeculectomy. Mitomycin-C was used under the conjunctival flap for up to 4 minutes (0,3mg/mL) and rinsed with 30mL saline solution. Scleral flap with crescent bevel and sclerectomy with a punch. Iridectomy and flap suture with nylon 10-0. Conjunctival suture with nylon 10-0.

Follow up after surgery was in the 1st, 4th, 7th, 15th, 30th days and after that monthly or whenever needed for clinical reasons.

ELIGIBILITY:
Inclusion Criteria:

* Patients with open angle glaucoma and uncontrolled IOP despite the use of maximum tolerated glaucoma medication.
* Patients over 18 years old.
* Patients who can understand and sign the inform consent form.

Exclusion Criteria:

* Other forms of glaucoma other than open angle glaucoma; previous psiquiatric condition ;
* Patients who can understand and sign the inform consent form;
* visual acuity worse than hand motion;
* previous retina surgery with buckle implant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-01; Primary Completion 2008-04 (Actual); Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
intra ocular pressure | Monthly

SECONDARY OUTCOMES:
number of hypotensive medications | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Paranhos JR, PHD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Gedde SJ, Schiffman JC, Feuer WJ, Parrish RK 2nd, Heuer DK, Brandt JD; Tube Versus Trabeculectomy Study Group. The tube versus trabeculectomy study: design and baseline characteristics of study patients. Am J Ophthalmol. 2005 Aug;140(2):275-87. doi: 10.1016/j.ajo.2005.03.031. PMID 16086949
- [Background] Minckler DS, Vedula SS, Li TJ, Mathew MC, Ayyala RS, Francis BA. Aqueous shunts for glaucoma. Cochrane Database Syst Rev. 2006 Apr 19;(2):CD004918. doi: 10.1002/14651858.CD004918.pub2. PMID 16625616
- [Result] Ishida K, Netland PA, Costa VP, Shiroma L, Khan B, Ahmed II. Comparison of polypropylene and silicone Ahmed Glaucoma Valves. Ophthalmology. 2006 Aug;113(8):1320-6. doi: 10.1016/j.ophtha.2006.04.020. PMID 16877071